CLINICAL TRIAL: NCT06439069
Title: BMI-Driven Tolerability and Efficacy of Entresto in Heart Failure Patients
Acronym: BETTER-HF
Status: Recruiting | Type: Observational
Sponsor: Lithuanian University of Health Sciences (Other)
Collaborators: Sligo General Hospital (Other); KlaipÄ-da University (Unknown)
Responsible Party: Principal Investigator, Ali Aldujeli, Consultant Cardiologist, Lithuanian University of Health Sciences
Other Study IDs: LUHSKC- 405
Record Dates: First submitted 2024-05-27; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure; Obesity
Keywords: Heart failure; Entresto; Obese; Sacubitril/Valsartan; BMI; Tolerability; Efficacy; NT-proBNP
MeSH Terms: conditions — Heart Failure; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (4):
- Normal Weight (BMI 18.5-24.9): Participants with a BMI between 18.5 and 24.9. This group will serve as a reference for normal weight individuals, providing baseline data for comparison with higher BMI categories regarding the tolerability and efficacy of Entresto.
- Overweight (BMI 25-29.9): Participants with a BMI between 25 and 29.9. This group will assess the impact of being overweight on the tolerability and efficacy of Entresto in heart failure patients.
- Obese (BMI 30-34.9): Participants with a BMI between 30 and 34.9. This group will evaluate the effects of obesity on the tolerability and efficacy of Entresto, providing insights into how increased body weight influences treatment outcomes.
- Very Obese (BMI ≥ 35): Participants with a BMI of 35 or higher. This group will explore the challenges and potential benefits of Entresto uptitration in very obese individuals, focusing on the highest BMI category.

SUMMARY:
This study aims to determine if patients with higher BMI can tolerate higher doses of Entresto (sacubitril/valsartan) and experience better symptomatic and functional outcomes compared to patients with lower BMI.

DETAILED DESCRIPTION:
This prospective cohort study will enroll heart failure patients with reduced ejection fraction (HFrEF) to evaluate the tolerability and efficacy of Entresto uptitration across different BMI categories (Normal weight, Overweight, Obese, and Very Obese). Primary outcomes include the maximum tolerable dose and incidence of adverse drug reactions. Secondary outcomes include changes in heart failure symptoms, functional capacity measured by the 6-minute walk test, hospitalization rates, and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and older
* Diagnosed with heart failure with reduced ejection fraction (HFrEF) (LVEF ≤ 35%)
* Naïve to Entresto therapy or willing to switch from previous ACE inhibitor/ARB therapy
* Ability to provide informed consent

Exclusion Criteria:

* Severe renal or hepatic impairment (e.g., eGFR < 30 mL/min/1.73m², severe liver disease)
* History of angioedema
* Pregnant or breastfeeding women
* Patients with malignancies or other severe comorbid conditions
* Non-compliance with medication regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study includes adult patients diagnosed with heart failure with reduced ejection fraction (HFrEF) and left ventricular ejection fraction (LVEF) ≤ 40%. Participants are either naïve to Entresto therapy or willing to switch from previous ACE inhibitor/ARB therapy. They will be categorized into four BMI groups: Normal Weight (BMI 18.5-24.9), Overweight (BMI 25-29.9), Obese (BMI 30-34.9), and Very Obese (BMI ≥ 35). Exclusion criteria include severe renal (eGFR < 30 mL/min/1.73m²) or hepatic impairment, history of angioedema, pregnancy, breastfeeding, active malignancies, severe comorbid conditions, and non-compliance with medication regimens. The study aims to enroll approximately 340 participants, with about 85 in each BMI category. Participants will be recruited from multiple cardiology clinics and hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerable dose of Entresto achieved | up to 24 weeks
  This outcome measures the highest dose of Entresto that patients in each BMI category can tolerate without experiencing significant adverse drug reactions (ADRs). The dose will be recorded at the end of the titration period, which is expected to last up to 24 weeks.

SECONDARY OUTCOMES:
Changes in Heart Failure Symptoms (NYHA Classification) | up to 24 weeks
  This outcome assesses the changes in heart failure symptoms based on the New York Heart Association (NYHA) classification at baseline and at 1 year follow-up visit. Improvement or worsening of symptoms will be tracked.
Changes in Functional Capacity (6-Minute Walk Test Distance) | up to 24 weeks
  This outcome measures the distance walked during the 6-minute walk test (6MWT) at baseline and at 1 year follow-up visit. It evaluates the functional capacity and exercise tolerance of participants.
Changes in Quality of Life (KCCQ Score) | up to 24 weeks
  This outcome assesses changes in the quality of life related to heart failure symptoms, as measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ). Scores will be recorded at baseline and at 1 year follow-up visit.
Hospitalization Rates | up to 24 weeks
  This outcome tracks the number of hospitalizations due to heart failure or related conditions during the study period. It provides an indicator of disease progression and treatment efficacy.
Changes in BNP/NT-proBNP Levels | up to 24 weeks
  This outcome measures the changes in B-type natriuretic peptide (BNP) or N-terminal pro b-type natriuretic peptide (NT-proBNP) levels, which are biomarkers for heart failure severity, at baseline and at 1 year follow-up visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided